CLINICAL TRIAL: NCT00253526
Title: Phase II Randomized Study of Surgical Resection and Adjuvant Gemcitabine Hydrochloride With Versus Without Bevacizumab in Patients With Adenocarcinoma of the Pancreas
Brief Title: Gemcitabine Hydrochloride With or Without Bevacizumab in Treating Patients Who Are Undergoing Surgery for Pancreatic Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000448825; NCI-05-C-0158; NCI-P6503; NCT00158392 (obsolete NCT alias)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2006-12

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage I Pancreatic Cancer; Stage II Pancreatic Cancer; Stage III Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Gemcitabine; Chemotherapy, Adjuvant; Immunization, Passive; Biological Therapy; Drug Therapy; Antibodies, Monoclonal; Surgical Procedures, Operative

INTERVENTIONS:
Drug: bevacizumab
Drug: gemcitabine hydrochloride
Procedure: adjuvant therapy
Procedure: anti-cytokine therapy
Procedure: antiangiogenesis therapy
Procedure: antibody therapy
Procedure: biological therapy
Procedure: chemotherapy
Procedure: conventional surgery
Procedure: growth factor antagonist therapy
Procedure: monoclonal antibody therapy
Procedure: surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells an help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of pancreatic cancer by blocking blood flow to the tumor. Giving gemcitabine hydrochloride together with bevacizumab after surgery may kill any remaining tumor cells.

PURPOSE: This phase II trial is studying gemcitabine hydrochloride and bevacizumab to see how well they work compared to gemcitabine hydrochloride alone in treating patients who are undergoing surgery for pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the disease-free interval in patients with adenocarcinoma of the pancreas treated with surgical resection followed by adjuvant gemcitabine hydrochloride with vs without bevacizumab.

Secondary

* Compare overall survival in patients treated with these regimens.
* Evaluate tumor gene expression profiles and levels of tumor angiogenesis markers to establish prognostic indicators for response in patients treated with these regimens.

OUTLINE: This is a randomized, controlled study.

All patients undergo surgical resection for the pancreatic tumor. Within 4-8 weeks after surgery, patients are stratified according to projected 2-year survival (≤ 5% vs > 5% and ≤ 33% vs > 33%). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride IV over 100 minutes on days 1, 8, and 15, and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for 6 courses. Patients then receive bevacizumab IV alone every 2 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive gemcitabine hydrochloride IV over 100 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 130 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas
* No evidence of distant metastasis on laparoscopy
* No superior mesenteric artery or thrombosed superior mesenteric vein involvement
* Superior mesenteric vein or portal vein involvement allowed
* Evidence of a pancreatic mass by radiographic or endoscopic examination

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 2,500/mm^3
* Absolute neutrophil count ≥ 1,250/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Hepatitis B surface antigen negative
* Hepatitis C virus negative
* No history of hepatic cirrhosis

Renal

* Creatinine ≤ 2.0 mg/dL
* Proteinuria negative or trace by urinalysis OR
* Protein < 1 g on 24 hr urine collection
* No active gross hematuria

Cardiovascular

* No severe congestive heart failure
* No active ischemic heart disease
* No ischemic changes on a cardiac thallium stress test
* No uncontrolled hypertension (i.e., blood pressure ≤ 150/100 mm Hg despite antihypertensive therapy)
* No active coagulation disorder

Pulmonary

* No active gross hemoptysis

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during the adjuvant therapy part of trial
* HIV negative
* No active infection
* No wound healing problem from recent invasive procedure
* No significant history of medical illness that would preclude patient from undergoing an operative procedure
* No other malignancy requiring systemic therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Recovered from prior immunotherapy for pancreatic cancer
* No prior bevacizumab

Chemotherapy

* Recovered from prior chemotherapy for pancreatic cancer
* No prior gemcitabine hydrochloride

Endocrine therapy

* Recovered from prior hormonal therapy for pancreatic cancer

Radiotherapy

* Recovered from prior radiotherapy for pancreatic cancer
* No prior radiotherapy to the pancreas

Surgery

* No prior definitive resection of the primary pancreatic tumor
* Prior surgery, other than resection of the primary tumor, allowed

Other

* More than 3 weeks since prior systemic therapy for this cancer
* No concurrent therapeutic anticoagulation causing elevated PT or PTT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Royal, MD, FACS, Principal Investigator — National Cancer Institute (NCI)